CLINICAL TRIAL: NCT04041310
Title: A Phase I/II, Multicenter, Open-Label Study of Nous-209 Genetic Vaccine for the Treatment of Microsatellite Unstable Solid Tumors
Brief Title: Nous-209 Genetic Vaccine for the Treatment of Microsatellite Unstable Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nouscom SRL (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOUS-209-01; IND #018954 (Other: FDA); 2021-002823-40 (EudraCT Number); MK-3475-E58 (Other: Merck Sharp & Dohme LLC); KEYNOTE-E58 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2019-07-21; First posted 2019-08-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor, Adult
Keywords: unresectable or metastatic dMMR tumor; MSI-H CRC; gastric tumor; gastro-esophageal junction (G-E junction) tumor
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase I. Part 1. Main Study of 26 weeks. Cohort A - Dose escalation. Cohort B - Expansion Cohort at RP2D Phase I. Part 2. Extended Follow-up week 27 to 110 in Cohorts A and B. Phase II: Expansion at RP2D of Nous-209 vaccine plus pembrolizumab combination therapy in adult subjects.
  * Cohort C (Phase II) - Subjects will be randomized with an allocation ratio 2:1 to Nous-209 vaccine plus pembrolizumab combination therapy versus pembrolizumab monotherapy.
  * Cohort D (Phase II) - Subjects who have had radiographic progression (PD) after having a best response of stable disease (SD) or better on/after anti-PD1 treatment.
  * In Phase I: 21 to 34 subjects will be enrolled across Cohorts A and B.
  * In Phase II: Cohort C: up to approximately 63 subjects, Cohort D: up to approximately 18 subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A - Dose-escalation (Experimental): Phase I. Part 1. Dose escalation cohort. Subjects treated with low dose or with high dose of GAd20-209-FSP prime and MVA-209-FSP boosts to define the RP2D, in combination with pembrolizumab.
  Phase I. Part 2 - Extended Follow-up from week 27 to week 110. Subjects with unresectable or metastatic deficient mismatch repair (dMMR) or MSI-H CRC, gastric, or gastro-esophageal junction (G-E junction) tumors.
  Interventions: Biological: GAd-209-FSP low dose; Biological: MVA-209-FSP low dose; Drug: KEYTRUDA®
- Cohort B - Expansion Cohort Phase I (Experimental): Phase I. Part 1. Expansion cohort at RP2D. Subjects treated with RP2D dose of GAd20-209-FSP prime and MVA-209-FSP boosts, in combination with pembrolizumab.
  Phase I. Part 2 - Extended Follow-up from week 27 to week 110. Subjects with unresectable or metastatic dMMR or MSI-H CRC, gastric, or G-E junction tumors.
  Interventions: Biological: GAd-209-FSP high dose; Biological: MVA-209-FSP high dose; Drug: KEYTRUDA®
- Cohort C - Expansion cohort Phase II (Experimental): Phase II. Subjects with locally advanced unresectable or metastatic, microsatellite instability high (MSI-H) or dMMR CRC who are eligible for anti-PD-1 1st line of treatment. Subjects will be randomized with an allocation ratio 2:1 to Nous-209 vaccine plus Keytruda® (pembrolizumab) combination therapy versus pembrolizumab monotherapy.
  Interventions: Biological: GAd20-209-FSP, RP2D; Biological: MVA-209-FSP, RP2D; Drug: KEYTRUDA®
- Cohort D - Expansion cohort Phase II (Experimental): Phase II. Subjects with locally advanced unresectable or metastatic, microsatellite instability high (MSI-H) or dMMR CRC who have had radiographic progression (PD) after having a best response of stable disease (SD) or better on/after anti-PD1 treatment. Nous-209 vaccine plus Keytruda® (pembrolizumab) combination therapy.
  Interventions: Biological: GAd20-209-FSP, RP2D; Biological: MVA-209-FSP, RP2D; Drug: KEYTRUDA®

INTERVENTIONS:
Biological: GAd-209-FSP low dose — GAd20-209-FSP IP, low dose
  Arms: Cohort A - Dose-escalation
Biological: MVA-209-FSP low dose — MVA-209-FSP IP, low dose
  Arms: Cohort A - Dose-escalation
Biological: GAd-209-FSP high dose — GAd20-209-FSP IP, high dose
  Arms: Cohort B - Expansion Cohort Phase I
Biological: MVA-209-FSP high dose — MVA-209-FSP IP, high dose
  Arms: Cohort B - Expansion Cohort Phase I
Biological: GAd20-209-FSP, RP2D — GAd20-209-FSP IP, RP2D
  Arms: Cohort C - Expansion cohort Phase II; Cohort D - Expansion cohort Phase II
Biological: MVA-209-FSP, RP2D — MVA-209-FSP IP, RP2D
  Arms: Cohort C - Expansion cohort Phase II; Cohort D - Expansion cohort Phase II
Drug: KEYTRUDA® — anti-PD-1 checkpoint inhibitor (200 mg; Q3W)
  Other Names: pembrolizumab

SUMMARY:
Ref: Protocol Version 9.1 05 December 2024. NOUS-209-01 is a multicenter, open-label, multiple cohorts, clinical study, designed to evaluate safety, tolerability, and immunogenicity, and to detect any preliminary evidence of anti-tumor activity of Nous-209 genetic polyvalent vaccine plus pembrolizumab combination therapy in adult subjects with unresectable or metastatic deficient mismatch repair (dMMR) or MSI-H CRC, gastric, or gastro-esophageal junction (G-E junction) tumors. Nous-209 is based on a heterologous prime/boost regimen composed of the Great Ape Adenovirus GAd20-209-FSP used for priming and Modified Vaccinia virus Ankara MVA-209-FSP used for boosting. The Phase I portion of the study is a first-in-human (FIH) clinical study with a primary objective to elucidate the safety and tolerability of Nous-209 in addition to establishing the recommended Phase 2 dose (RP2D), whereas the Phase II was introduced to assess efficacy as the primary objective.

DETAILED DESCRIPTION:
Ref: Protocol Version 9.1 05 December 2024. Both Frame Shift Peptide (FSP) neoantigen-encoding genetic vaccines are administered intramuscularly using 1 prime with the GAd20-209-FSP and 3 boosts with MVA-209-FSP in combination with Keytruda®, the licensed programmed death receptor-1 (PD-1)-blocking antibody pembrolizumab, in adult subjects with unresectable or metastatic Mismatch Repair Deficient (dMMR) or MSI-H colorectal cancer (CRC), gastric, or G-E junction tumors. In Phase I, GAd20-209-FSP prime will be administered on the day of 2nd pembrolizumab infusion (week 4); MVA-209-FSP boosts will be administered on the day of 3rd, 4th and 5th pembrolizumab infusion (weeks 7 and 10 and 13). In Phase II, GAd20-209-FSP prime will be administered on the same day as the 1st pembrolizumab infusion (day 1, week 1); MVA-209-FSP boosts will be administered in week 2 and at the time of the 2nd and 3rd pembrolizumab infusions (weeks 4 and 7).

The study is composed of a Phase I divided in two parts and a Phase II, as described below :

Phase I:

* Cohort A - Dose escalation Cohort of Nous-209 vaccine plus pembrolizumab combination therapy in adult subjects with unresectable or metastatic deficient mismatch repair (dMMR) or MSI-H CRC, gastric, or gastro-esophageal junction (G-E junction) tumors;
* Cohort B - Expansion Cohort at Recommended Phase 2 Dose (RP2D) of Nous-209 vaccine plus pembrolizumab combination therapy in adult subjects with unresectable or metastatic dMMR or MSI-H CRC, gastric, or G-E junction tumors. Part 2 - Extended Follow-up from week 27 to week 110.

Phase I (Cohorts A and B): The Sponsor estimates that the trial will require approximately 24 months from the time the first subject signs the informed consent until the last subject's last visit at week 26 (Main Study); and approximately 42 months until last subject's last visit at week 110 (Extended follow up).

Phase II:

Expansion at RP2D of Nous-209 vaccine plus Keytruda® (pembrolizumab) combination therapy in adult subjects in the following study population:

* Cohort C (Phase II) - Subjects with locally advanced unresectable or metastatic, microsatellite instability high (MSI-H) or dMMR CRC who are eligible for anti-PD-1 1st line of treatment. Subjects will be randomized with an allocation ratio 2:1 to Nous-209 vaccine plus pembrolizumab combination therapy versus pembrolizumab monotherapy.
* Cohort D (Phase II) - Subjects with locally advanced unresectable or metastatic, microsatellite instability high (MSI-H) or dMMR CRC who have had radiographic progression (PD) after having a best response of stable disease (SD) or better on/after anti-PD1 treatment.

Phase II (Cohorts C and D): Participation duration per subject is expected to last up to 18 months in Cohort C and up to 12 months in Cohort D.

Subjects who do not progress might stay in extended follow-up for up to approximately 2 years (106 weeks or completion of 35 administrations of pembrolizumab).

Enrollment in Phase I and II is now terminated.

ELIGIBILITY:
Inclusion Criteria for Cohort C (Phase II)

In order to be eligible, the subject must:

1. Have the ability to comprehend and willingness to provide written informed consent (ICF) for the study.
2. Have previously proven microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) status (confirmatory testing is not required);

   • dMMR/MSI Testing: Patients are eligible to the combined treatment based on previous diagnosis for dMMR/MSI status. dMMR/MSI status diagnosis should be performed locally by IHC or NGS or PCR based tests that are certified per local requirementss (Hara et al. 2018; Boland et al. 1998) CDx ™, 2017.
3. Patients with locally advanced unresectable or metastatic, microsatellite instability high (MSI-H) or mismatch repair deficient (dMMR) CRC who are eligible for anti-PD-1 1st line of treatment.
4. Be ≥18 years of age on day of signing informed consent.
5. Have a life expectancy of at least 6 months.
6. Have a performance status of 0 - 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
7. Have resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 2 or less (except alopecia). If subject received major surgery or radiation therapy they must have recovered from the toxicity and/or complications from the intervention.
8. Have adequate organ function as defined in the following tables (Table 1. Adequate Organ Function Laboratory Values ). Specimens must be collected within 10 days prior to the start of study treatment. If any hematological or chemistry values are outside the specified range during the initial screening, rescreening process may be conducted to reassess and ensure compliance with the adequate organ function criteria as outlined in Table 1.
9. Not be previously treated with a (licensed or experimental) anti-PD-1 or anti-PD-L1 checkpoint inhibitor.
10. If participating in translational reasearch [see Section 7.0.6 Translational research (only selected sites)], agree to have a biopsy at baseline from a lesion that can be biopsied with an acceptable clinical risk (as judged by the Investigator in discussion with the interventional radiologist or endoscopist). An older (not older than 6 months) FFPE specimen from locations not radiated prior to biopsy can be accepted. Furthermore, optionally agree to have another biopsy taken on-treatment if not representing an unacceptable clinical risk and/or if technically feasible as judged by the Investigator in discussion with the interventional radiologist or endoscopist.
11. Have measurable disease per RECIST version 1.1.
12. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
13. Females: not be pregnant (see Appendix 7: Contraceptive Guidance and Pregnancy Testing), not breastfeed, and must have at least one of the following conditions that apply:

    • Not a woman of childbearing potential (WOCBP) as defined in Appendix 7: Contraceptive Guidance and Pregnancy Testing OR

    • A WOCBP who agrees to use highly effective contraceptive methods as outlined in Appendix 7: Contraceptive Guidance and Pregnancy Testing during the treatment period and for at least 180 days after the last dose of study treatment and refrain from egg donation during this period.
14. Fertile male patients: agree to use a contraceptive as detailed in Appendix 7:

Contraceptive Guidance and Pregnancy Testing of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.

Inclusion Criteria for Cohort D (Phase II):

In order to be eligible, the subject must:

1. Have the ability to comprehend and willingness to provide written informed consent (ICF) for the study.
2. Have previously proven microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) status (confirmatory testing is not required); dMMR/MSI Testing: Patients are eligible to the combined treatment based on previous diagnosis for dMMR/MSI status. dMMR/MSI status diagnosis should be performed locally, by IHC or NGS or PCR based tests that are certified per local requirements (Hara et al. 2018; Boland et al. 1998) CDx ™, 2017.
3. Patients with locally advanced unresectable or metastatic MSI-H/dMMR CRC who have had radiographic progression (PD) after having a best response of stable disease (SD) or better on/after anti-PD-1 treatment.
4. May have progressed on additional approved therapy.
5. Be ≥18 years of age on day of signing informed consent.
6. Have a life expectancy of at least 6 months.
7. Have a performance status of 0 - 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
8. Have resolution of toxic effect(s) of the most recent prior cancer therapies to Grade 2 or less (except alopecia). If patient received major surgery or radiation therapy they must have recovered from the toxicity and/or complications from the intervention.
9. Have adequate hematological and blood chemistry values for Phase II as indicated in Table 1. Adequate Organ Function Laboratory Values. The specimens must be collected within 10 days prior to the start of study treatment. If any hematological or chemistry values are outside the specified range during the initial screening, rescreening process may be conducted to reassess and ensure adequate organ function criteria as outlined in Table 1.
10. If participating in translational research [see Section 7.0.6 Translational research (only selected sites)], agree to have a biopsy at baseline from a lesion that can be biopsied with an acceptable clinical risk (as judged by the Investigator in discussion with the interventional radiologist or endoscopist). An older (not older than 6 months) FFPE specimen from locations not radiated prior to biopsy can be accepted.

    Furthermore, optionally agree to have another biopsy taken on-treatment if not representing an unacceptable clinical risk and/or if technically feasible as judged by the Investigator in discussion with the interventional radiologist or endoscopist.
11. Have measurable disease per RECIST version 1.1.
12. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
13. Females: not be pregnant (see Appendix 7: Contraceptive Guidance and Pregnancy Testing), not breastfeed, and must have at least one of the following conditions that apply:

    • Not a woman of childbearing potential (WOCBP) as defined in Appendix 7: Contraceptive Guidance and Pregnancy Testing OR

    • A WOCBP who agrees to use highly effective contraceptive methods as outlined in Appendix 7: Contraceptive Guidance and Pregnancy Testing during the treatment period and for at least 180 days after the last dose of study treatment and refrain from egg donation during this period.
14. Male patients: agree to use a contraceptive as detailed in Appendix 7: Contraceptive Guidance and Pregnancy Testing of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.

Table 1: Adequate Organ Function Laboratory Values

Hematological

* Absolute neutrophil count (ANC) ≥1500/µL
* Platelets ≥100 000/µL
* Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (1)

Renal Creatinine OR Measured or calculated creatinine (2) clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR

* 30 mL/min for participant with creatinine levels >1.5 × institutional ULN

Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

Coagulation [Optional]

* International normalized ratio (INR) OR prothrombin time (PT)
* Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT)= alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)= aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR= glomerular filtration rate; ULN= upper limit of normal.

1. Criteria must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Participants can be on stable dose of erythropoietin (≥ approximately 3 months).
2. Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria for Cohort C and D (Phase II)

The patient must be excluded from participating in if he/she:

1. Has a diagnosis of immunodeficiency, or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
2. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (have no evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any worsening of neurologic symptoms with respect to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to pembrolizumab.
3. Is expected to require any form of systemic or localized antineoplastic therapy while on study other than the study drugs.

   • Phase IIa and Cohort C only: Had prior adjuvant treatment with an anti-PD1, or PD-L1 or PD-L2 agent or an antibody targeting other immunoregulatory receptors or mechanisms.
4. Cohort D only:

   • discontinued prior therapy with a checkpoint inhibitor due to Grade 3, or higher, treatment-related toxicities.
5. Had prior allogeinic tissue or solid organ transplant.
6. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
7. Has known history of HIV (HIV1/2 antibodies). HIV-infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

   1. Participants on ART must have a CD4+ T-cell count >350 cells/mm3 at time of screening
   2. Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening.
   3. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (Day 1)
8. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
9. Had prior radiotherapy within 2 weeks of enrollment, or within 4 weeks of enrollment in the case of radiation to central nervous system (CNS), which requires

   ≥4-week washout. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. Note: A one-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) for non-CNS disease.
10. Has immunosuppression implying the continued use of systemic (at prednisone dose equivalent of >10 mg) or topical steroids, at or near, the planned intramuscular injection site or the use of immunosuppressive agents for any concurrent condition in the 4 weeks prior to first study treatment administration. Inhaled and eye dropcontaining corticosteroids are permitted.
11. Has received a live-virus vaccination within 30 days of pembrolizumab start. Seasonal flu vaccines that do not contain live virus are permitted. Covid-19 vaccines are permitted under the following guidance: mRNA Covid-19 vaccines are permitted if administered more than 2 weeks prior to Study Day 1, and Covid19 Adenovirusbased vaccines are accepted if administrated at least 6 months before Study Day 1.

    Administration of killed vaccines are allowed.
12. Has an active severe infection requiring therapy.
13. Has active HBV or HCV infection that requires treatment, or at risk for HBV reactivation (i.e., positive hepatitis B surface antigen [HBsAg]). Patients with negative HBsAg and positive total hepatitis B core antibody may be included if HBV DNA is undetectable at the time of screening. Patients who are positive for HCV antibody are eligible only if the PCR test is negative for HCV RNA. Patients with known current or prior HBV infection must have HBsAg and HBV DNA testing during screening and those with current or previous HCV infection must have HCV DNA testing.
14. Has a chronic illness including, but not limited to, chronic heart failure, coronary heart disease, cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Has any history of anaphylaxis in reaction to a vaccination.
16. Is a woman who is pregnant or breastfeeding.
17. Any condition in the judgment of the Investigator, which makes the patient unsuitable for study participation; including psychological condition.
18. Has known hypersensitivity to pembrolizumab or to components of the Nous-209 study therapy or its analogues (including a known history of allergy to egg proteins).
19. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease

      ≥5 years before the first dose of study treatment and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease.
20. Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 4 weeks prior to first dose of study treatment or concurrent enrolment in another clinical study.
21. Has active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
22. Is receiving growth factors including, but not limited to, granulocyte colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, etc., within 4 weeks of study drug administration.

Revaccination Eligibility Criteria for participants receiving Nous-209 with pembrolizumab (Phase II) All participants that have been treated with Nous-209 and pembrolizumab combination in Phase IIa and in Phase IIb (Cohorts C and D) will be offered revaccination with Nous209 approximately 6 months after starting treatment (Table 3: Schedule of Activities for revaccination of eligible patients in Phase IIa and Phase IIb (Cohorts C and D)) providing the following criteria are met:

1. Being in objective radiological stable disease according to RECIST v1.1 without any prior evidence of Partial response (PR), complete response (CR), or progressive disease (PD), based on the last available on-treatment scan prior to revaccination.
2. Have no limiting toxicities preventing further administration of pembrolizumab (see Appendix 4: Management of Immune-Related Adverse Events).
3. Continues to fufil the eligibility criteria for enrolment, except for the following inclusion criterion of Cohort C participants:

   •9. Not have been previously treated with a (licensed or experimental) anti-PD1 or anti-PD-L1 checkpoint inhibitor.
4. Revaccination is not permitted for patients in Phase IIb Cohort C receiving pembrolizumab only.
5. Participants who meet the criteria for revaccination may only receive revaccination once. During the revaccination period, participants will receive the same prime-boost vaccination doses and regimen of GAd20-209 FSP and MVA-209-FSP as in the original vaccination treatment period. Participants will continue to receive pembrolizumab at 200 mg Q3W.

Image acquisitions and tumour assessments should continue on their regular imaging schedule for the duration of treatment (see Section 7.1 Schedule of Activities (SoA) (Phase II)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Toxicity (DLT assessment), in Phase I, Cohort A | Within 28 days
  Toxicity analyzed within 28-days from the administration of the prime vaccination with GAd20-209-FSP
Safety and Tolerability, in Phase I, Cohort A and B. | Up to 110 weeks
  AEs as characterized by type, severity (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v.5.0), timing, seriousness, and relationship to study treatments.
Overall Response Rate (ORR) at any time during the study, in Phase II (Cohort C and D). | 18 months
  Assessed using RECIST v1.1

SECONDARY OUTCOMES:
Immunogenicity (T cell responses against vaccine FSPs) in Phase I, Cohorts A and B | Through study completion, an average of 2 years
  PBMC-derived T cell responses against vaccine FSPs, as measured by IFN-gamma ELISpot
Safety and tolerability (local and systemic AEs), in Phase II (Cohort C and D) | Up to 18 months
  AEs as characterized by type, severity (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v.5.0), timing, seriousness, and relationship to study treatments. Assessed by standard using RECIST v1.1 criteria at 6, 12 and 18 months.

OTHER OUTCOMES:
Clinical: Overall Response Rate (ORR), in Phase I, Cohort A and B | Phase I Main Study and Extended follow-up. Up to 110 weeks
  Assessed by tumor imaging using RECIST v1.1
Clinical: Disease Control Rate (DCR), in Phase I, Cohort A and B | Phase I Main Study and Extended follow-up. Up to 110 weeks
  Assessed by tumor imaging using RECIST v1.1
Clinical: Time to Tumor Response (TTR), Phase I Main Study and Extended follow-up. | Phase I Main Study and Extended follow-up. Up to 110 weeks.
  Assessed by the Investigator using RECIST v1.1, and Overall Survival (OS)
Clinical: Duration of Response (DoR), Phase I Main Study and Extended follow-up, Phase II (Cohost C and D) | Up to 110 weeks
  Assessed by tumor imaging using RECIST v1.1
Clinical: Progression-free survival (PFS), Phase I Main Study and Extended follow-up, Phase II (Cohort C and D) | Up to 110 weeks
  Assessed by tumor imaging using RECIST v1.1
Clinical: Overall Survival (OS), Phase I Main Study and Extended follow-up. | Up to 110 weeks
  Assessed by tumor imaging using RECIST v1.1
Clinical: Best Overall Response (BOR), Phase II (Cohort C and D). | Up to 18 months
  Assessed by tumor imaging using RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sven Gogov, MD, Study Director — Nouscom SRL
Locations (46):
- United States (13):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Comprehensive Cancer Center, Irvine, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Newport Beach, California
  - Mt. Sinai, Miami Beach, Florida
  - Boca Raton Clinical Research, Plantation, Florida
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, Division of Oncology, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medicine / New York-Presbyterian Hospital, New York, New York
  - MD Anderson Cancer Center (MDACC), Houston, Texas
- Belgium (3):
  - Cliniques Universitaires Saint-Luc - Centre du Cancer, Brussels
  - Centre Hospitalier de l'Ardenne - Libramont - Clinique du Sein, Libramont
  - CHU de Liège, Liège
- Canada (2):
  - Mount Sinai Hospital, Toronto
  - Princess Margaret Cancer Center, Toronto
- Italy (6):
  - Aorn Sg Moscati, Avellino
  - Candiolo cancer Center,FPO IRCCS, Candiolo
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale Niguarda, Milan
  - AOUS Policlinico Le Scotte, Siena
- Spain (21):
  - Hospital Universitario de A Coruna, A Coruña
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia Hospitalet, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Asistencial de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital General Universitario de Valencia, Valencia
  - University Clinical Hospital Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- University College London Hospitals NHS Foundation Trust Cancer Clinical Trials Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Non-clinical results published by D'Alise (Nouscom Srl) et al. in Nature Communications — https://www.ncbi.nlm.nih.gov/pubmed/31217437